CLINICAL TRIAL: NCT04877886
Title: A Novel Technique for the Assessment of Non-traumatic Pain Diagnosis in the Emergency Department.
Brief Title: TCHCCT-Zhong-Xing-Emergency-Department Ultrasound With IV Contrast in Acute Flank Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Hung,Tzu-Yao, Emergency Medicine Physician, Taipei City Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: TCHCCT-ZXERUSC
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Acute Flank Pain
Keywords: Acute flank pain; Ultrasound; IV contrast
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ultrasound with IV contrast (Experimental): use ultrasound with IV contrast to perform in acute flank pain patient
  Interventions: Diagnostic Test: Ultrasound with IV contrast
- CT with IV contrast (Active Comparator): to compare with ultrasound with IV contrast in acute flank pain patient
  Interventions: Diagnostic Test: CT with IV contrast
- Ultrasound without IV contrast (Active Comparator): baseline for the Ultrasound with IV contrast
  Interventions: Diagnostic Test: Ultrasound without IV contrast
- CT without IV contrast (Active Comparator): baseline for the CT with IV contrast
  Interventions: Diagnostic Test: CT without IV contrast

INTERVENTIONS:
Diagnostic Test: Ultrasound with IV contrast — To compare the efficiency over the ultrasound scan within contrast
  Arms: Ultrasound with IV contrast
Diagnostic Test: CT with IV contrast — CT with IV contrast
  Arms: CT with IV contrast
Diagnostic Test: Ultrasound without IV contrast — Ultrasound without IV contrast
  Arms: Ultrasound without IV contrast
Diagnostic Test: CT without IV contrast — CT without IV contrast
  Arms: CT without IV contrast

SUMMARY:
To evaluate the efficiency of ultrasound with IV contrast and compare this with the Computed Tomography in acute flank pain patient at Emergency Department.

DETAILED DESCRIPTION:
Acute flank pain is a common chief complaint in emergency departments (ED), but it is a challenge for physicians in ED to accurately diagnose. It can cause variable diseases and is in many cases lethal (e.g. aortic dissection, ruptured aortic aneurysm, renal artery dissection, ruptured tumor, etc). The computed tomography scan with IV contrast is an ideal tool to diagnose due to its high sensitivity and specificity and is a golden standard examination. However, currently point-of-care ultrasound is routinely used as first-line technique. As this procedure is non-invasive and has no radiative effect, it is considered more logical, especially for those critical patients who are not able to move and perform the CT scan. Furthermore, the iodine contrast of CT scan is known as renal toxicity and should be used with caution in patient with hyperthyroidism and allergy to the contrast. The radiation of CT scan would be harmful to the pregnant patient as well.

IV contrast ultrasound is a novel technique nowadays and it is widely used in diagnosing breast, liver, renal and pancreatic tumors. The ultrasound contrast using air microbubbles could enhance the scanning quality and also has high sensitivity and specificity. In ED, ultrasound with contrast now could be applied to the abdominal trauma and pediatric injury. For those patients with poor renal function, thyroid disease and pregnant women who cannot undergo IV contrast CT, IV contrast ultrasound provides a faster and safer way to evaluate patients in ED. We compared CT and ultrasound with IV contrast to determine the difference in efficiency between both examinations.

ELIGIBILITY:
Inclusion Criteria:

* Acute flank pain who visit ER

Exclusion Criteria:

* Younger than 18 years old
* Known allergy to contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic rate of ultrasound with IV contrast in acute flank pain patient | The hospitalization of each participant, up to 28 days
  Evaluate the sensitivity and specificity in ultrasound scan

SECONDARY OUTCOMES:
To compare the efficiency over the ultrasound and CT scan within or without contrast | The hospitalization of each participant, up to 28 days
  compared the sensitivity and specificity between CT and ultrasound scan

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Yao Hung, MD, Study Director — Taipei City Hospital ZhongXing Branch
Locations (1):
- Taipei City Hospital Zhong-Xing branch, Taipei, Taiwan